CLINICAL TRIAL: NCT00410904
Title: Phase 2 Study of AZD2171 (NSC 732208) in Combination With Pemetrexed in Relapsed Non-Small Cell Lung Cancer (NOS: 10029514)
Brief Title: AZD2171 and Pemetrexed Disodium in Treating Patients With Relapsed Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00165; NCI-2009-00165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000517316; 2006-042 (Other: Wayne State University/Karmanos Cancer Institute); 7389 (Other: CTEP); P30CA022453 (NIH); U01CA062487 (NIH)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Recurrent Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cediranib; Pemetrexed

ARMS (1):
- Arm I (Experimental): Patients receive oral AZD2171 once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: cediranib maleate
  Other Names: AZD2171; Recentin
Drug: pemetrexed disodium
  Other Names: ALIMTA; LY231514; MTA

SUMMARY:
This phase II trial is studying how well giving AZD2171 together with pemetrexed disodium works in treating patients with relapsed non-small cell lung cancer. AZD2171 and pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. AZD2171 may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving AZD2171 together with pemetrexed disodium may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the response rate in patients with relapsed non-small cell lung cancer treated with AZD2171 and pemetrexed disodium.

SECONDARY OBJECTIVES:

I. Assess the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to prior bevacizumab treatment (yes vs no).

Patients receive oral AZD2171 once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks* in the absence of disease progression or unacceptable toxicity.

[Note: * The first course is 4 weeks in duration; all subsequent courses are 3 weeks in duration.]

After completion of study treatment, patients are followed at 4 weeks and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* Lesions in a previously irradiated area are considered measurable provided there has been an increase of >= 10 mm since completion of radiotherapy
* Received 1-2 prior regimens, including 1 doublet chemotherapy regimen, AND meets 1 of the following criteria:

  * No prior bevacizumab (cohort A)
  * Patients with squamous cell carcinoma, treated and controlled brain metastases, or history of hemoptysis allowed
* Received 1-2 prior regimens*, including 1 doublet chemotherapy regimen, AND meets 1 of the following criteria:

  * Previously treated with bevacizumab (cohort B)
  * No discontinuation of bevacizumab for uncontrollable hypertension and/or life-threatening bleeding
  * Must have disease progression after prior bevacizumab (NOTE: *Prior adjuvant therapy is considered 1 regimen if disease progression occurred within 1 year of completion of therapy; if a regimen was discontinued within 2 courses for allergic reaction or unacceptable drug-specific toxicity, that regimen dose not count)
* No large pleural effusion or ascites unless drained
* No active brain metastases by brain MRI or CT scan within the past 4 weeks
* Patients with treated, controlled brain metastasis allowed provided they are neurologically stable without seizures within the past 3 weeks
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* WBC >= 3,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 2.5 times ULN (< 5 times ULN if liver metastases present)
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Urine protein =< 1+ on 2 consecutive dipsticks taken >= 1 week apart
* No significant hemorrhage (i.e., > 30 mL in 1 episode) within the past 3 months
* No significant hemoptysis (i.e., > 5 mL fresh blood in 1 episode) within the past 4 weeks
* No active gastrointestinal disease that may affect the ability of the patient to absorb AZD2171
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171 or pemetrexed disodium
* No other malignancies within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would preclude study compliance
* No New York Heart Association class III or IV heart disease
* Mean QTc < 470 msec by ECG
* No history of familial long QT syndrome
* Fertile patients must use effective contraception
* No resting blood pressure (BP) consistently > 140/90 mm Hg; Patients whose BP is controlled after starting, adjusting, or increasing medication allowed
* LVEF normal by MUGA or echocardiogram for patients at increased risk for left ventricular dysfunction, as evidenced by any of the following:

  * Prior treatment with anthracyclines
  * New York Heart Association class III or IV heart disease or controlled class II disease
  * Prior central thoracic radiotherapy, including radiotherapy to the heart
  * Myocardial infarction within the past 12 months
* At least 4 weeks since prior definitive chest radiotherapy (> 60 Gy) and recovered
* At least 3 months since prior craniotomy for resection of brain metastasis
* At least 3 weeks since prior radiotherapy for brain metastases
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 2 weeks since prior palliative radiotherapy
* At least 2 weeks since prior surgery (excluding the placement of vascular access or drainage of pleural effusion or ascites) and recovered
* No inability or unwillingness to take folic acid, cyanocobalamin (vitamin B12), or dexamethasone
* No prior pemetrexed disodium
* At least 5 half-lives since prior and no concurrent drugs or biologics with proarrythmic potential including:

  * Amiodarone hydrochloride
  * Arsenic trioxide
  * Bepridil
  * Chloroquine
  * Chlorpromazine
  * Cisapride
  * Clarithromycin
  * Disopyramide
  * Dofetilide
  * Domperidone
  * Droperidol
  * Erythromycin
  * Halofantrine
  * Haloperidol
  * Ibutilide
  * Mesoridazine
  * Methadone
  * Pentamidine
  * Pimozide
  * Procainamide
  * Sotalol
  * Sparfloxacin
  * Thioridazine
* Not pregnant or nursing
* More than 30 days since prior investigational agents and recovered
* No aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) for 2 days before, during, and for 2 days after pemetrexed disodium administration: Low-dose aspirin (≤ 325 mg/day) for vascular disorders allowed
* No long-acting NSAIDs (e.g., naproxen, piroxicam, diflunisal, nabumetone, or celecoxib) for 5 days before, during, and for 2 days after pemetrexed disodium
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No other concurrent investigational agents
* Life expectancy > 12 weeks
* No concurrent medications that can markedly affect renal function (e.g., vancomycin or amphotericin)
* Negative pregnancy test
* Relapsed disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirish Gadgeel, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic.
Groups:
- Arm I Cohort A- No Prior Bevacizumab (Avastin); Arm I Cohort B- Prior Bevacizumab (Avastin): Patients receive oral AZD2171 30 mg orally once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium 500mg/m2 IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I Cohort A- No Prior Bevacizumab (Avastin) | Arm I Cohort B- Prior Bevacizumab (Avastin)
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I Cohort A- No Prior Bevacizumab (Avastin); Arm I Cohort B - Prior Bevacizumab (Avastin): Patients receive AZD2171, 30 mg orally once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium 500mg/m2 in 100 ml of 0.9% sodium chloride, IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm I Cohort A- No Prior Bevacizumab (Avastin) | Arm I Cohort B - Prior Bevacizumab (Avastin) | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Median (Full Range); unit: years] | 61 (8.342) [44 to 79] | 58.5 (9.101) [39 to 78] | 59.5 (8.5683686) [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 21 | 10 | 31
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial) 2 Separate Cohorts of Relapsed NSCLC Cohort A: Pts Who Have Received Prior Chemo w/o Ever Having Received Bevacizumab. Cohort B: Pts Who Have Received Prior Bevacizumab.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v 1.0) for target lesions and assessed by MRI or CT:
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  Overall Response (OR) = CR + PR, the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started)
Time Frame: Up to 4 years
Measure: Number; unit: participants
Groups:
- Arm I - Cohort A, no Prior Bevacizumab (Avastin); Arm I - Cohort B, Prior Bevacizumab (Avastin): Patients receive oral AZD2171 30 mg orally once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium 500mg/m2 IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I - Cohort A, no Prior Bevacizumab (Avastin) | Arm I - Cohort B, Prior Bevacizumab (Avastin)
Number analyzed (Participants) | 40 | 20
participants | 10 | 4

2. Secondary Outcome: Progression-free Survival
Description: Estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates of all PFS and OS statistics will be calculated. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: The duration of time from start of treatment to time of progression, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I: Patients receive oral AZD2171 once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  cediranib maleate
  pemetrexed disodium
Arm/Group | Arm I
Number analyzed (Participants) | 60
months | 5.6 [4.1 to 6.8]

3. Secondary Outcome: Overall Survival
Description: Estimated with the standard Kaplan-Meier method, from which summary statistics of interest (median, 1-year rate, etc.) will be derived. Both point and 95% confidence interval estimates of all PFS and OS statistics will be calculated.
Time Frame: The time from start of treatment to time of death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 60
months | 11.5 [6.9 to 14.0]

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of treatment
Groups:
- Arm I - Cohort A: This is a one arm study with two cohorts.
  Cohort A: No prior bevacizumab before entering into this trial
  Patients receive AZD2171, 30 mg orally once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium 500mg/m2 in 100 ml of 0.9% sodium chloride, IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
- Arm I - Cohort B: This is a one arm study with two cohorts.
  Cohort B: Prior bevacizumab before entering into this trial
  Patients receive AZD2171, 30 mg orally once daily on days 1-28 in course 1 and on days 1-21 in course 2 and all subsequent courses. Patients also receive pemetrexed disodium 500mg/m2 in 100 ml of 0.9% sodium chloride, IV over 10 minutes on day 8 in course 1 and on day 1 in course 2 and all subsequent courses. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I - Cohort A | Arm I - Cohort B
Serious Adverse Events (participants affected / at risk) | 7/40 | 2/20
Other Adverse Events (participants affected / at risk) | 33/40 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Cohort A (N=40) | Arm I - Cohort B (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Death NOS (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PROGRESSION OF NSCLC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CNS CEREBROVASCULAR ISCHEMIA (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Cohort A (N=40) | Arm I - Cohort B (N=20)
Anemia (Blood and lymphatic system disorders) | 19 (19) | 11 (11)
Hypothyroidism (Endocrine disorders) | 9 (9) | 5 (5)
ABDOMINAL CRAMPING (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 16 (16) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 28 (28) | 16 (16)
Flatulence (Gastrointestinal disorders) | 4 (4) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (22) | 10 (10)
Oral pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 11 (11) | 6 (6)
Edema limbs (General disorders) | 5 (5) | 4 (4)
Fatigue (General disorders) | 33 (33) | 18 (18)
Pain (General disorders) | 3 (3) | 5 (5)
Upper respiratory infection (Infections and infestations) | 7 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (8) | 4 (4)
Alanine aminotransferase increased (Investigations) | 17 (17) | 8 (8)
Alkaline phosphatase increased (Investigations) | 6 (6) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 12 (12) | 8 (8)
Creatinine increased (Investigations) | 11 (11) | 3 (3)
INCREASED BUN (Investigations) | 2 (2) | 3 (3)
Lymphocyte count decreased (Investigations) | 7 (7) | 2 (2)
Neutrophil count decreased (Investigations) | 12 (12) | 11 (11)
Platelet count decreased (Investigations) | 20 (20) | 10 (10)
Weight loss (Investigations) | 9 (9) | 8 (8)
White blood cell decreased (Investigations) | 22 (22) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 27 (27) | 15 (15)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 29 (29) | 20 (20)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (17) | 10 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 6 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 21 (21) | 11 (11)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Pemetrexed was approved for front line therapy based on the results of a phase III study; it became known that pemetrexed is ineffective in pts.with squamous cell lung ca. It was also challenging to combine VEGF-TKIS with chemo this pt. population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less